CLINICAL TRIAL: NCT00164151
Title: A Comparison of the Efficacy and Safety of Two Bowel Preparations: HalfLytely® (2L NuLYTELY and 20 mg Bisacodyl), and Visicol™ Prior To Colonoscopy.
Brief Title: A Comparison of the Efficacy and Safety of HalfLytely Vs Visicol Prior To Colonoscopy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: F38-23
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Colonoscopy
Keywords: colonoscopy preparation; prep

INTERVENTIONS:
Drug: HalfLytely
Drug: Visicol

SUMMARY:
The objective of this study is to determine the efficacy and safety of HalfLytely as compared to Visicol as bowel preparations before colonoscopic examination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for routinely accepted indications, Evaluation of BE results, GI bleeding, Anemia of unknown etiology, Neoplastic disease surveillance, Endosonography, Inflammatory bowel disease (except as noted below), Unknown diarrhea etiology, Polypectomy, Laser therapy, Foreign body removal and decompression (except as noted below).
* 18 years of age or older.
* Otherwise in good health, as determined by physical exam and medical history.
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, or vasectomized spouse).
* Subjects with electrolyte abnormalities such as hypernatremia, hyperphosphatemia, hypokalemia, or hypocalcemia must have them corrected prior to study participation.
* Subject has read and signed the written informed consent document prior to study participation.

Exclusion Criteria:

* Subjects with known or suspected bowel perforation or obstruction, severe inflammatory bowel disease, ileus, acute alimentary tract surgery, significant gastroparesis or gastric outlet obstruction, appendicitis, gastric retention, toxic colitis, toxic megacolon, or massive and/or abnormal rectal bleeding.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects with uncontrolled cardiovascular disease.
* Subjects with congestive heart failure.
* Subjects with unstable angina pectoris.
* Subjects with ascites.
* Subjects with renal insufficiency.
* Subjects who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days.
* Subjects who are pregnant or lactating.
* Subjects who are allergic to polyethyleneglycol.
* Subjects who are allergic to sodium phosphate salts.
* Subjects who are currently taking, or plan to take, other sodium phosphate- containing products, such as enemas or non-prescription liquid purgatives.
* Subjects with pre-existing electrolyte disturbances, such as dehydration, or those secondary to the use of diuretics.
* Subjects who are taking drugs that may affect electrolyte levels.
* Subjects receiving non-study laxatives, antacids and prokinetic agents during the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-06; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Bowel preparation success: preparation rated as "good" or "excellent" by the blinded investigator.

SECONDARY OUTCOMES:
Safety: review of preparation symptoms, adverse events and laboratory testing.
Patient acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brady, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- San Antonio, Texas, United States